CLINICAL TRIAL: NCT00269477
Title: Persistence of Bactericidal Antibodies in Adolescents and Adults Aged 15 to 23 Years Who Received a Single Dose of Menactra® or Menomune®-A/C/Y/W-135 Five Years Earlier
Brief Title: Persistence of Antibodies in Adolescents and Adults 15 to 23 Years Who Received One Dose of Menactra® or Menomune®
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA35
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Results first posted 2009-12-14 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Meningitis; Meningococcal Infection
Keywords: Meningitis; Meningococcal infection; Neisseria meningitidis; Menactra®; Menomune®
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Menactra® Vaccine Group 1 (Experimental): Participants had previously received a dose of Menactra® vaccine in Study MTA02,did not participate in Study MTA19 (NCT 00777790). They provided a pre-vaccination blood sample on Day 0, received one booster dose of Menactra® vaccine on Day 0 and provided 3 additional blood samples on Day 3, Day 7, and Day 28 post-vaccination.
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Menactra® Vaccine Group 2 (Experimental): Participants had previously received a dose of Menactra® vaccine in Study MTA02,did not participate in Study MTA19 (NCT 00777790). They provided a pre-vaccination blood sample on Day 0, received one booster dose of Menactra® vaccine on Day 0 and provided 3 additional blood samples on Day 5, Day 14, and Day 28 post-vaccination
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Meningococcal Vaccine-naive Group 3 (Active Comparator): Participants have never received Meningococcal vaccine and provided one blood sample pre-vaccination on Day 0, received a dose of Menactra® vaccine on Day 0, and provided 3 additional blood samples on Day 3, Day 7, and Day 28 post-vaccination.
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Meningococcal Vaccine-naive Group 4 (Active Comparator): Participants have never received Meningococcal vaccine and provided one blood sample pre-vaccination on Day 0, received a dose of Menactra® vaccine on Day 0, and provided 3 additional blood samples on Day 5, Day 14, and Day 28 post-vaccination.
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Vaccine Group 1
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Vaccine Group 2
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Meningococcal Vaccine-naive Group 3
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Meningococcal Vaccine-naive Group 4

SUMMARY:
The study is designed to evaluate the persistence of bactericidal antibodies in subjects aged 15 to 23 years (not yet 24 years) who had been vaccinated five years previously in Study MTA02 and did not participate in Study MTA19 (NCT 00777790). In addition, the kinetics of the antibody response will be evaluated in a subset of these participants who will receive a booster dose of Menactra® vaccine. This will be compared to aged matched control subjects who have not been previously vaccinated with a meningococcal vaccine or had documented meningitis disease who will also receive a dose of Menactra® vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy, as determined by medical history.
* Subject is between the ages of 15 and 23 years (not yet 24 years).
* For subjects who participated in Study MTA02, subject previously received one dose of Menactra® vaccine or Menomune®-A/C/Y/W-135 vaccine.
* Did not participate in Study MTA19 (a subset of subjects from Study MTA02 who had been recruited for a follow-up challenge study)
* Subject or parent/legal guardian has signed an Institutional Review Board (IRB)-approved informed consent form and subject has signed an IRB-approved assent form.
* Before recruitment for the second part of the study, subjects should be thoroughly screened to ensure that they are able to comply with protocol specifications
* A negative urine pregnancy test is required for menstruating female subjects.

Exclusion Criteria:

* History of documented invasive meningococcal disease.
* Received any other meningococcal vaccine
* Received any vaccine (other than desensitization therapy for allergies) in the 28-day period prior to enrollment
* Scheduled to receive any vaccination in the 28-day period after enrollment
* Received systemic antibiotic therapy within the 72 hours prior to collection of a blood sample
* Actively enrolled or scheduled to be enrolled in another clinical study
* Serious chronic disease (i.e., cardiac, renal, neurologic, rheumatologic, metabolic, gastrointestinal, hematologic, psychiatric, or other organ system)
* Known or suspected impairment of immunologic function
* Acute medical illness with or without fever within 72 hours or an oral temperature ≥ 100.4°F (≥ 38.0°C) at the time of inclusion
* Administration of immune globulin, other blood products, or corticosteroid within 3 months of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Personal or family history of Guillain-Barre Syndrome
* Suspected or known hypersensitivity to any of the vaccine components
* Unavailable for the entire study period or unable to attend the scheduled visits or to comply with the study procedures
* Any condition, which in the opinion of the investigator would pose a health risk to the participant.

Ages: 15 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 145 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (8):
- United States (8):
  - Atlanta, Georgia
  - Marietta, Georgia
  - Woburn, Massachusetts
  - Akron, Ohio
  - Columbus, Ohio
  - Sellersville, Pennsylvania
  - Kingsport, Tennessee
  - Norfolk, Virginia

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 20 December 2005 to 31 May 2006, in 8 United States clinical sites.
Pre-assignment Details: A total of 145 participants who participated in a previous study MTA02 and other meningococcal-vaccine naive participants were enrolled.
Groups:
- Menactra® Vaccine Group 1: Participants had previously received a dose of Menactra® vaccine in Study MTA02,did not participate in Study MTA19 (NCT 00777790). They provided a pre-vaccination blood sample on Day 0, received one booster dose of Menactra vaccine on Day 0 and provided 3 additional blood samples on Day 3, Day 7, and Day 28 post-vaccination.
- Menactra® Vaccine Group 2: Participants had previously received a dose of Menactra® vaccine in Study MTA02,did not participate in Study MTA19 (NCT 00777790). They provided a pre-vaccination blood sample on Day 0, received one booster dose of Menactra vaccine on Day 0 and provided 3 additional blood samples on Day 5, Day 14, and Day 28 post-vaccination.
- Meningococcal Vaccine-naive Group 3: Participants have never received Meningococcal vaccine and provided one blood sample pre-vaccination on Day 0, received a dose of Menactra vaccine on Day 0, and provided 3 additional blood samples on Day 3, Day 7, and Day 28 post-vaccination
- Meningococcal Vaccine-naive Group 4: Participants have never received Meningococcal vaccine and provided one blood sample pre-vaccination on Day 0, received a dose of Menactra vaccine on Day 0, and provided 3 additional blood samples on Day 5, Day 14, and Day 28 post-vaccination.
Period: Overall Study
Arm/Group | Menactra® Vaccine Group 1 | Menactra® Vaccine Group 2 | Meningococcal Vaccine-naive Group 3 | Meningococcal Vaccine-naive Group 4
Started | 9 | 18 | 58 | 60
Completed | 4 | 12 | 57 | 60
Not Completed | 5 | 6 | 1 | 0
Not completed — Protocol Violation | 5 | 5 | 1 | 0
Not completed — Missed post-vaccination blood draw | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Vaccine Group 1 | Menactra® Vaccine Group 2 | Meningococcal Vaccine-naive Group 3 | Meningococcal Vaccine-naive Group 4 | Total
Number analyzed (Participants) | 9 | 18 | 58 | 60 | 145
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 10 | 53 | 54 | 122
  Between 18 and 65 years | 4 | 8 | 5 | 6 | 23
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.1 (1.62) | 18.8 (1.86) | 16.4 (1.38) | 16.6 (1.81) | 17.9 (2.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 13 | 27 | 28 | 73
  Male | 4 | 5 | 31 | 32 | 72
Region of Enrollment [Number; unit: participants]
  United States | 9 | 18 | 58 | 60 | 145

OUTCOME MEASURES:

1. Primary Outcome: Participants With Serum Bactericidal Activity of ≥ 1:8 for Each Menactra® Vaccine Serogroups Pre-vaccination and 28 Days Post-booster or Post-primary Dose Vaccination.
Description: Groups 1 and 2 received booster vaccination, Groups 3 and 4 received primary vaccination.
  Serum bactericidal activity for each Menactra® vaccine serogroups were at pre-vaccination and at 28 days post-booster or post-primary vaccination.
Time Frame: 28 days post-vaccination (5 years after Menactra® or Menomune® vaccination)
Population: SBA-BR titer for each of the 4 meningococcal serogroups in the vaccine was evaluated in the per-protocol population.
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group 1 | Menactra® Vaccine Group 2 | Meningococcal Vaccine-naive Group 3 | Meningococcal Vaccine-naive Group 4
Number analyzed (Participants) | 4 | 12 | 57 | 60
Participants
  Meningococcal serogroup A - Day 0 | 4 | 12 | 25 | 25
  Meningococcal serogroup A - Day 28 | 4 [1677.5 to 320034.7] | 12 [14221.4 to 47563.3] | 56 [15101.3 to 29164.0] | 60 [12672.1 to 26079.6]
  Meningococcal serogroup C - Day 0 | 2 | 8 | 15 | 20
  Meningococcal serogroup C - Day 28 | 4 [2803.6 to 191496.7] | 12 [8654.7 to 62032.2] | 56 [4405.0 to 11319.3] | 60 [3472.0 to 8413.3]
  Meningococcal serogroup Y - Day 0 | 3 | 12 | 49 | 52
  Meningococcal serogroup Y - Day 28 | 4 [161.4 to 294032.5] | 12 [5353.8 to 31586.0] | 57 [3453.0 to 7346.6] | 60 [2833.2 to 5921.5]
  Meningococcal serogroup W-135 - Day 0 | 3 | 12 | 25 | 28
  Meningococcal serogroup W-135 - Day 28 | 4 [5578.8 to 96234.1] | 12 [7461.5 to 50878.1] | 57 [6158.1 to 14240.4] | 60 [5178.0 to 10773.2]

2. Other Pre Specified Outcome: Number of Participants Reporting Solicited Injection Site and Solicited Systemic Reactions
Description: Solicited injection site reactions: Erythema, Swelling, and Pain. Solicited systemic reactions: Fever (temperature), Headache, Malaise, and Myalgia.
Time Frame: Day 0 to 7 post-vaccination
Population: Safety analysis was on all enrolled and vaccinated participants, intend-to-treat population
Measure: Number; unit: Participants
Arm/Group | Menactra® Vaccine Group 1 | Menactra® Vaccine Group 2 | Meningococcal Vaccine-naive Group 3 | Meningococcal Vaccine-naive Group 4
Number analyzed (Participants) | 9 | 18 | 58 | 60
Participants
  Any Erythema | 2 | 2 | 13 | 14
  Grade 3 Erythema (≥ 2 inches) | 1 | 0 | 1 | 0
  Any Swelling | 1 | 0 | 12 | 3
  Grade 3 Swelling (≥ 2 inches) | 1 | 0 | 1 | 0
  Any Injection Site Pain | 2 | 8 | 36 | 37
  Grade 3 Injection Site Pain (Incapacitating) | 0 | 0 | 0 | 0
  Any Fever | 0 | 0 | 2 | 0
  Grade 3 Fever (≥ 39.6 ºC) | 0 | 0 | 0 | 0
  Any Headache | 0 | 5 | 20 | 28
  Grade 3 Headache (Prevents daily activities) | 0 | 1 | 0 | 1
  Any Malaise | 1 | 3 | 15 | 22
  Grade 3 Malaise (Prevents daily activities) | 0 | 0 | 0 | 0
  Any Myalgia | 2 | 6 | 24 | 28
  Grade 3 Myalgia (Prevents daily activities) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 28 days post-booster or post-primary Menactra® vaccination
Arm/Group | Menactra® Vaccine Group 1 | Menactra® Vaccine Group 2 | Meningococcal Vaccine-naive Group 3 | Meningococcal Vaccine-naive Group 4
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/18 | 0/58 | 0/60
Other Adverse Events (participants affected / at risk) | 1/9 | 5/18 | 32/58 | 23/60
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Vaccine Group 1 (N=9) | Menactra® Vaccine Group 2 (N=18) | Meningococcal Vaccine-naive Group 3 (N=58) | Meningococcal Vaccine-naive Group 4 (N=60)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3)
Injection site induration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Venipuncture site bruise (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 4 (4) | 3 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 6 (6) | 1 (1)
Joint sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 9 (9) | 11 (18)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (3) | 2 (2) | 2 (4) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 3 (4)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.